CLINICAL TRIAL: NCT00166660
Title: Preterm Fetal Growth Restriction and Developmental Care
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Heidelise Als, PhD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD046855 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-03

CONDITIONS: Preterm Birth
Keywords: Preterm infants; Developmental Care; NIDCAP; Fetal Growth Restriction; Neurobehavior; APIB; MRI; EEG; Parent Stress
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: NIDCAP (Newborn Individualized Developmental Care) — The NIDCAP model aims to create a relationship-based developmentally supportive care environment for the preterm infant and family. The theory proposes that care implementation that takes into account the infants' thresholds of disorganization is most supportive of long term outcome. Specifically, the intervention consisted of weekly neurobehavioral observations and reports of the experimental group infants' behavior with suggestions for parents and staff in ways to support each infant's development. The developmental specialists formally observed each infant's behavior weekly throughout the hospitalization, starting with the phase of the infant's initial stabilization, and then every seven days throughout hospital discharge and to 2wCA.

SUMMARY:
The goal of the project is to show the effectiveness of individualized developmental care and intervention, which begins with the FGR preterm infant's admission to the newborn intensive care unit (NICU) and extends to 2 weeks (w) after full term equivalent age or 2w CA (corrected age for prematurity).

DETAILED DESCRIPTION:
The protocol aims to demonstrate the effectiveness of an intervention geared to significantly improve functional competence for preterm infants with fetal growth restriction (FGR). Incidence of FGR is estimated to be as high as 5% of the general obstetric population. Preterms with FGR are doubly jeopardized. Aside from much higher mortality rates they also show significantly increased morbidity rates, including significant learning disabilities and school failure (>50%). The intervention's underlying premise holds that it is far more effective to support the immature brain, which is compromised by FGR, to develop optimally before the infant reaches full term rather than to attempt to ameliorate increasingly deviant development after deviance has occurred. The goal of the project is to show the effectiveness of individualized developmental care and intervention, which begins with the FGR preterm infant's admission to the newborn intensive care unit (NICU) and extends to 2 weeks (w) after full term equivalent age or 2w CA (corrected age for prematurity). Intervention in the NICU is considered more advantageous for the infant's later development than delay of intervention until after discharge home. The proposal maintains that the last trimester of gestation is a critical period for brain development, especially when compromised by FGR. In-NICU intervention at this critical brain development time is expected to reduce the infants' hypersensitivity and reactivity while in the NICU, and to lead to reduction of the high incidence of behavioral problems in infancy, which frequently foreshadows later behavioral and learning problems as well as school failure.

The study aims to test three related hypotheses:

1. Individualized developmental NICU care and intervention will enhance FGR preterm infants' brain development both functionally and structurally.
2. The in-NICU intervention will improve the parents' understanding of their infant's individuality and equip them to feel more competent as parents.
3. The intervention itself, while individualized for each infant, will be quantifiable and reliably reproducible.

The study will:

1. Test the effectiveness of the intervention by assessing brain development and functional adaptation of a high risk preterm population (n=30) with documented intrauterine FGR and born between 28 and 33w gestational age.
2. Assess the FGR preterm infants' neurodevelopment within one week from birth (baseline) and again at 2w CA (outcome).
3. Compare the results on the effectiveness of the intervention for the FGR preterm infants to a recently studied cohort of appropriately grown (AGA) preterm infants born at comparable gestational ages, supported with the same intervention and measured in comparable ways.

The primary infant measures proposed will be brain functional (EEG coherence, neurobehavioral functioning) and brain structural assessments (MRI). The goal will be to examine the direct causal connections and correlations among population characteristics, the intervention, and ultimate outcome at 2w CA. The project is expected to deliver comprehensive and substantive results in favor of the developmental NICU intervention for FGR preterm infants as well as for the earlier studied AGA population. The proposed study is expected to demonstrate intervention effectiveness in improving FGR preterm infants' neurodevelopment. It is anticipated that the intervention-based improvement in brain structure and function will set the stage for improvement in later performance, especially in terms of behavioral/emotional adaptation, learning and school achievement, which are all critical for life success.

ELIGIBILITY:
Inclusion Criteria:

* Inborn at Brigham and Women's Hospital, Boston
* Gestational age ≥28 and ≤33 weeks
* Doppler diagnosed absent or reversed end-diastolic umbilical artery flow velocity
* Less than 5th percentile in birthweight and head circumference for gestational age

Exclusion Criteria:

* Major chromosomal or congenital anomalies
* Major congenital infections
* Significant prenatal diagnosed focal brain lesions
* Uncontrolled maternal illness
* History of smoking, alcoholism, and use of illicit drugs
* History of significant maternal deprivation, abuse, or malnutrition
* No telephone access and/or insufficient English language facility

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2004-07; Primary Completion 2008-12 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of Preterm Infants' Behavior (APIB) | 2 weeks corrected age (2w CA)
Quantified Electroencephalography (qEEG) | 2 weeks Corrected Age (2w CA)
Magnetic Resonance Imaging(MRI) | 2 weeks Corrected Age (2w CA)

SECONDARY OUTCOMES:
Parent Stress Level | 2 weeks Corrected Age (2w CA)

CONTACTS AND LOCATIONS:
Overall Officials: Heidelise Als, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts

REFERENCES:
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237